CLINICAL TRIAL: NCT03871179
Title: Cognoa ASD Diagnostic Device - Data Collection Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Cognoa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1189568
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Masking Description: Participants, care providers, and diagnostic clinicians are blinded to the diagnostic output of the ASD diagnostic device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ASD Diagnostic Device (Other): The ASD Diagnostic Device is a machine learning algorithm-based software as a medical device that is incorporated into a parent/caregiver-facing mobile application, the "Cognoa App", used outside of a clinical setting
  Interventions: Diagnostic Test: ASD Diagnostic Device

INTERVENTIONS:
Diagnostic Test: ASD Diagnostic Device — The ASD Diagnostic Device is a machine learning algorithm-based software as a medical device that is incorporated into a parent/caregiver-facing mobile application, the "Cognoa App", used outside of a clinical setting

SUMMARY:
The primary objective of this study is to collect data to ascertain the PPV and NPV of the current version of the Cognoa diagnostic device. A secondary objective is to collect data, in the form of additional questions, in order to train new algorithms related to children's developmental and behavioral conditions.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 months of age and < 72 months of age
* Functional English capability in the home environment
* Documented parental and/or clinician concern for developmental delay
* Participants must have a smartphone capable of downloading the Cognoa App (Cognoa supports iOS 10.0 and up, Android 6.0 and up)

Exclusion Criteria:

* Children with suspected auditory or visual hallucinations or with prior diagnosis of childhood onset schizophrenia.
* Children with known sensory impairment such as deafness or blindness
* Children with known physical impairment affecting their ability to use their hands
* Children with major dysmorphic features or prenatal exposure to teratogens (such as fetal alcohol syndrome)
* Children with history or diagnosis of genetic conditions (such as Rett's syndrome or fragile X)
* Children with microcephaly
* Children with history or prior diagnosis of epilepsy or seizures
* Children with history of or suspected neglect
* Children with history of brain defect, injury or insult requiring interventions such as surgery or chronic medication
* Children whose age on the date of enrollment is outside the target age range
* Children who have been previously enrolled in any Cognoa clinical study or survey
* Children whose medical records had been included in any internal Cognoa training or validation sets

Ages: 18 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Positive and negative predictive value of ASD Dx in relation to clinician diagnostic evaluation | approximately one month

CONTACTS AND LOCATIONS:
Overall Officials: Tom Megerian, MD, Principal Investigator — Children's Hospital of Orange County
Locations (1):
- Children's Hospital of Orange County, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol